CLINICAL TRIAL: NCT06621680
Title: Effect of Connective Tissue Massage on Premenstrual Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Enas Nabil Georgy, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005312
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Geritol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multivitamins group (Active Comparator): This group will receive multivitamins capsule once daily, for 12 weeks.
  Interventions: Drug: Multivitamins
- Connective tissue massage group (Experimental): This group will receive multivitamins in addition to connective tissue massage on (Sacral, lumbar, last thoracic vertebrae-T12, and subcostal regions), 2 sessions/week, 20 minutes/ session for 12 weeks
  Interventions: Drug: Multivitamins; Other: Connective tissue massage

INTERVENTIONS:
Drug: Multivitamins — All participants will receive multivitamins (vitatron) capsule once daily, for 12 weeks.
Other: Connective tissue massage — Connective tissue massage will be applied on (Sacral, lumbar, last thoracic vertebrae-T12, and subcostal regions), 2 sessions/week for 20 minutes each session for 12 weeks. Treatment will begin 3 days before menstruation to the 4th day of menstruation for 3 successive menstrual cycles.
  Arms: Connective tissue massage group

SUMMARY:
This study will be conducted to investigate the effect of connective tissue massage on premenstrual syndrome.

DETAILED DESCRIPTION:
Premenstrual syndrome is a collection of emotional, physiological and behavioral symptoms that develop around the end of the luteal phase and fade away with or after mensturation.

The physiological effects of connective tissue massage (CTM) are both local and general. Local effects include release of histamine from mast cells which leads to a triple response, local swelling and arteriolar dilatation mediated by local axon reflexes. The increased blood flow to the region assists resolution of subacute or chronic inflammation and reduces pain by removing nocigenic chemicals from the tissues. The mechanical distortions produced by CTM strokes help to mobilize connective tissue and improve function.

Few studies have investigated the effect of the CTM on premenstrual syndrome in adolescent females. So this study will be conducted to add new information about the effect of connective tissue massage on premenstrual syndrome, which may help adolescent females suffering from this syndrome in decreasing their symptoms, thus adding new information to the field of physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Virgin adolescent females diagnosed with premenstrual syndrome.
* Their age will be ranged from 17-25 years (3 years post puberty).
* Their body mass index (BMI) will be less than 30 kg/m2 .
* All are of regular menstrual cycles.
* All of them suffering from moderate and severe PMS.

Exclusion Criteria:

Participants will be excluded from this study if they have

* Any pathological finding in the pelvic cavity as polycystic ovarian syndrome, endometriosis, and pelvic inflammatory diseases.
* Irregular menstruation.
* Any history of gynecological intervention.
* Open wounds, weak/broken bones or fractures.

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 3 months
  Degrees of menstrual pain will be assessed using a VAS for all participants before and after treatment, which is a method of representing pain on a 10 cm linear scale.
  A score of zero means "No pain" and 10 means "a very high degree of pain".
Premenstrual syndrome severity | 3 months
  Severity of premenstrual symptoms will be assessed by using the Menstrual Distress Questionnaire (MDQ). Each participant will examine symptom categories (pain, concentration, water retention, behavior changes, negative effect, autonomic reaction, arousal and control) Participants are asked to report the symptoms experienced during their most recent menstrual period, using a rating scale. Responses ranged from (0) No experience of the symptom, (1) mild, (2) moderate, (3) severe and (4) very severe disabling symptoms. Overall scores are interpreted as follows: >50- mild, 50 to 70- moderate and >70 severe

CONTACTS AND LOCATIONS:
Overall Officials: Azza B Kassab, professor, Study Chair — Cairo University
Locations (1):
- Enas Nabil Georgy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol